CLINICAL TRIAL: NCT07326072
Title: The Comparative Study of Electromagnetic Navigation Bronchoscopic With Ultra-thin Cryobiopsy and Forceps Biopsy in the Diagnosis of Peripheral Pulmonary Nodules
Brief Title: The Study of ENB With Ultra-thin Cryobiopsy in the Diagnosis of Peripheral Pulmonary Nodules
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MR-11-25-060861
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Diagnosis
Keywords: Diagnosis; Peripheral pulmonary lesions; Cryobiopsy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: The subjects were randomly (1:1) divided into groups. Cryobiopsy was assigned to the experimental group, while biopsy using a biopsy forceps was assigned to the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryobiopsy group (Experimental): Electromagnetic Navigation Bronchoscopic with Ultra-thin Cryobiopsy
  Interventions: Procedure: Cryobiopsy
- Forceps biopsy group (Active Comparator): Electromagnetic Navigation Bronchoscopic with Forceps Biopsy
  Interventions: Procedure: Forceps biopsy

INTERVENTIONS:
Procedure: Cryobiopsy — Cryobiopsy : Insert a 1.1mm cryoprobe along the electromagnetic navigation catheter, obtain samples with at least 2 pieces each.
  Arms: Cryobiopsy group
Procedure: Forceps biopsy — Forceps biopsy:Insert 1.8mm forceps along the electromagnetic navigation catheter, obtain at least five tissue samples through precise clamping.
  Arms: Forceps biopsy group

SUMMARY:
To investigate the safety and efficacy of ultrafine cryoprobe biopsy by electromagnetic navigation bronchoscopy compared with biopsy forceps in the diagnosis of peripheral pulmonary nodules in a national multicenter randomized controlled trial

DETAILED DESCRIPTION:
This project intends to carry out a national multicenter randomized controlled study, with traditional forceps biopsy as the control group and cryobiopsy as the experimental group, to verify the feasibility, effectiveness and safety of electromagnetic navigation bronchoscope-guided cryobiopsy in the diagnosis of peripheral pulmonary nodules, so as to provide an efficient and minimally invasive diagnostic method for the diagnosis of peripheral pulmonary nodules

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 90 years;
2. pulmonary nodules detected by chest CT, suspected malignant nodules or unknown cause should be confirmed by biopsy;
3. chest CT showed that the nodule was located in the segmental bronchus and below, and the maximum diameter of the nodule was 8 mm to 30 mm.It was not accessible by conventional bronchoscopy;
4. if chest CT showed multiple pulmonary nodules, one of the pulmonary nodules was selected as the target lesion.

Exclusion Criteria:

1. contraindications to the bronchoscopy procedure;
2. high risk of bleeding, such as bronchial artery penetration or suspected lung metastasis of renal cell carcinoma;
3. electromagnetic source implanted in the body;
4. contraindications to anesthesia;
5. pregnant woman;
6. participated in other studies within three months and did not withdraw or finish, affect the observation of this study;
7. inability or unwillingness to provide informed consent or comply with the follow-up schedule.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | follow-up for 12 months
  The primary outcome was the diagnostic yield of ENB-guided cryobiopsy and forceps biopsy for diagnosing pulmonary lesions

SECONDARY OUTCOMES:
Adverse events | follow-up for one month
  Adverse events related to the research

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Doctor, Study Chair — Beijing Chaoyang Hospital, China
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will share clinical date.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for sharing for 2 years after formal publication of the study.
Access Criteria: Researchers working on cryobiopsy and electromagnetic navigation bronchoscopy.

REFERENCES:
- [Result] Balasubramanian P, Abia-Trujillo D, Barrios-Ruiz A, Garza-Salas A, Koratala A, Chandra NC, Yu Lee-Mateus A, Labarca G, Fernandez-Bussy S. Diagnostic yield and safety of diagnostic techniques for pulmonary lesions: systematic review, meta-analysis and network meta-analysis. Eur Respir Rev. 2024 Sep 18;33(173):240046. doi: 10.1183/16000617.0046-2024. Print 2024 Jul. PMID 39293856
- [Result] Tang Y, Tian S, Chen H, Li X, Pu X, Zhang X, Zheng Y, Li Y, Huang H, Bai C. Transbronchial lung cryobiopsy for peripheral pulmonary lesions. A narrative review. Pulmonology. 2024 Sep-Oct;30(5):475-484. doi: 10.1016/j.pulmoe.2023.08.010. Epub 2023 Oct 31. PMID 37914556
- [Result] Bondue B, Schlossmacher P, Allou N, Gazaille V, Taton O, Gevenois PA, Vandergheynst F, Remmelink M, Leduc D. Trans-bronchial lung cryobiopsy in patients at high-risk of complications. BMC Pulm Med. 2021 Apr 26;21(1):135. doi: 10.1186/s12890-021-01503-9. PMID 33902504
- [Result] Matsumoto Y, Nakai T, Tanaka M, Imabayashi T, Tsuchida T, Ohe Y. Diagnostic Outcomes and Safety of Cryobiopsy Added to Conventional Sampling Methods: An Observational Study. Chest. 2021 Nov;160(5):1890-1901. doi: 10.1016/j.chest.2021.05.015. Epub 2021 May 19. PMID 34022184
- [Result] Nakai T, Watanabe T, Kaimi Y, Ogawa K, Matsumoto Y, Sawa K, Okamoto A, Sato K, Asai K, Matsumoto Y, Ohsawa M, Kawaguchi T. Safety profile and risk factors for bleeding in transbronchial cryobiopsy using a two-scope technique for peripheral pulmonary lesions. BMC Pulm Med. 2022 Jan 10;22(1):20. doi: 10.1186/s12890-021-01817-8. PMID 35000601
- [Result] Nakai T, Watanabe T, Kaimi Y, Shiomi K, Ando K, Miyamoto A, Ogawa K, Matsumoto Y, Sawa K, Sato K, Asai K, Matsumoto Y, Mikami Y, Ohsawa M, Kawaguchi T. Diagnostic Utility and Safety of Non-Intubated Cryobiopsy Technique Using a Novel Ultrathin Cryoprobe in Addition to Conventional Biopsy Techniques for Peripheral Pulmonary Lesions. Respiration. 2023;102(7):503-514. doi: 10.1159/000531010. Epub 2023 Jun 28. PMID 37379810
- [Result] Kim MH, Kim SH, Lee G, Mok J, Lee MK, Song JS, Eom JS. Next-generation sequencing using tissue specimen collected with a 1.1 mm-diameter cryoprobe in patients with lung cancer. Respirology. 2024 Apr;29(4):333-339. doi: 10.1111/resp.14680. Epub 2024 Feb 20. PMID 38379178
- [Result] Kim SH, Mok J, Kim S, Yoo WH, Jo EJ, Kim MH, Lee K, Kim KU, Park HK, Lee MK, Eom JS. Clinical outcomes of transbronchial cryobiopsy using a 1.1-mm diameter cryoprobe for peripheral lung lesions - A prospective pilot study. Respir Med. 2023 Oct;217:107338. doi: 10.1016/j.rmed.2023.107338. Epub 2023 Jun 26. PMID 37380091

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT07326072/Prot_SAP_002.pdf
  • Informed Consent Form (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT07326072/ICF_003.pdf